CLINICAL TRIAL: NCT00152256
Title: A Phase 3,6-Month, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Two Doses of Asoprisnil Versus Placebo in Subjects With Uterine Leiomyomata
Brief Title: A Study to Evaluate of the Safety and Effectiveness of Asoprisnil in Treating Women With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-037
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Fibroid Uterus; Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Fibroids
Keywords: Symptomatic Uterine Fibroids; Excessive Uterine Bleeding; Uterine Hemorrhage
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Metrorrhagia; Uterine Hemorrhage | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — Asoprisnil 10 mg Tablet, oral Daily for 6 months
  Other Names: J867
  Arms: 1
Drug: Asoprisnil — Asoprisnil 25mg Tablet, oral Daily for 6 months
  Other Names: J867
  Arms: 2
Drug: Placebo — Placebo Tablet, oral Daily for 6 months
  Arms: 3

SUMMARY:
The objective of this study is to determine the safety and efficacy effects of two doses of asoprisnil (10 mg and 25 mg) compared with placebo when administered daily for 6 months to premenopausal subjects with symptomatic uterine leiomyomata.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of abnormal uterine bleeding associated with uterine fibroids. Asoprisnil (10 mg and 25mg) is being evaluated in a Phase 3 program to establish long term safety and effectiveness and therefore provide women with a medical alternative to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* History of regular menstrual cycles (21-42 days)
* Diagnosis of uterine fibroid(s)
* Abnormal vaginal bleeding associated with uterine fibroids
* Otherwise in good health
* Subject must have at least one fibroid with a diameter ≥ 2 cm or multiple small fibroids with a uterine volume of ≥ 200 cm3

Exclusion Criteria:

* Less than 3 months postpartum and post-lactation
* Previous myomectomy within 1 year
* Any abnormal lab or procedure result the study-doctor considers important
* Severe reaction(s) to or are currently using any hormone therapy
* History of osteoporosis or other bone disease

Ages: 18 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2003-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Cumulative percent of subjects achieving amenorrhea. | Month 3

SECONDARY OUTCOMES:
Change from baseline in total symptom severity score and the Uterine Fibroid Symptom-Quality of Life total score. | Final Visit
Change from baseline in menorrhagia, metrorrhagia, bloating, pelvic pressure, dysmenorrhea, pelvic pain and urinary symptoms. | Final Visit
Change from baseline in the Work Limitation Questionnaire Index. | Final Visit
Change from baseline in the two dimensions of the SF-36 (Physical Component Summary and Mental Component Summary). | Final Visit
Change from baseline in the monthly bleeding score. | Final Visit
Change from baseline in the hemoglobin concentration. | Final Visit
Change from baseline in volume of the largest fibroid. | Final Visit
Percentage of subjects who discontinue with the intent to have surgery for fibroids during treatment. | During treatment period
Percentage of subjects who respond positively to the global efficacy question. | Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott